CLINICAL TRIAL: NCT05080283
Title: A Pre-Marketing, Prospective, Single-Site, Open-Label, Within-Subject, Actual-Use, Interventional Study of Acceptance and Performance With Experienced Adult Cochlear Implant Recipients Using the CP1110 Sound Processor Compared With the CP1000 Sound Processor
Brief Title: Acceptance and Performance of CP1110 Sound Processor With Experienced Adult Cochlear Implant Recipients.
Acronym: PINNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5810
Record Dates: First submitted 2021-09-19; First posted 2021-10-15 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-01

CONDITIONS: Adult Cochlear Implant Recipients
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Prospective, pre-market, single-site, non-randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CP1110 with automated ForwardFocus On (SCAN 2 FF), CP1110 with ForwardFocus Off (SCAN 2), and CP1000 (Other): All participants assigned to CP1110 Sound Processor System with automated ForwardFocus On (SCAN 2 FF), CP1110 Sound Processor System with ForwardFocus Off (SCAN 2) compared to the previously marketed Nucleus 7 Sound Processor (Model: CP1000) in a random order.
  Interventions: Device: CP1110 Sound Processor System with automated ForwardFocus On (SCAN 2 FF); Device: Nucleus 7 Sound Processor (model: CP1000) system; Device: CP1110 Sound Processor System with ForwardFocus Off (SCAN 2)

INTERVENTIONS:
Device: CP1110 Sound Processor System with automated ForwardFocus On (SCAN 2 FF) — Sound Processor
Device: Nucleus 7 Sound Processor (model: CP1000) system — Sound Processor
Device: CP1110 Sound Processor System with ForwardFocus Off (SCAN 2) — Sound Processor

SUMMARY:
The clinical study aims to investigate acceptance, actual-use usability and speech performance with a new behind-the-ear sound processor (model number: CP1110) system, compared with the commercially available Nucleus 7 Sound Processor (model: CP1000) system, with particular focus on the acceptance of and satisfaction with a noise reduction feature in the Automatic Scene Classifier 'SCAN 2'.

DETAILED DESCRIPTION:
The clinical study aims to investigate acceptance, actual-use usability and speech performance with a new behind-the-ear sound processor (model number: CP1110) system, compared with the commercially available Nucleus 7 Sound Processor (model: CP1000) system, with particular focus on the acceptance of and satisfaction with a noise reduction feature in the Automatic Scene Classifier 'SCAN 2'. This study will build on the evidence collected in previous Nucleus 7 Sound Processor take home studies and will also aim to confirm the in-booth performance of CP1110 and Nucleus 7 Sound Processors.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Post lingually deafened.
3. Implanted with the CI600 Series (CI612, CI632, CI622, CI624), CI500 Series (CI512, CI532, CI522) or Freedom Series (CI24RE(CA), CI24RE(ST), CI422).
4. At least 6 months experience with a cochlear implant.
5. At least 3 months experience with a Nucleus 7 (CP1000) Sound Processor
6. Able to score 30% or more at +15 SNR with CI alone on a sentence in babble test
7. Willingness to participate in and to comply with all requirements of the protocol.
8. Fluent speaker in English as determined by the investigator
9. Willing and able to provide written informed consent

Exclusion Criteria:

1. Additional disabilities that would prevent participation in evaluations.
2. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedures.
3. Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
4. Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
5. Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.
6. Currently participating, or participated in another interventional clinical study/trial in the past 30 days or if less than 30 days, the prior investigation was Cochlear sponsored and determined by the investigator to not impact clinical findings of this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cochlear Sydney, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nel E, Hong W, Playford J, Mashal ME. A clinical and real-world investigation of cochlear implant recipient speech performance in noise with the automation of ForwardFocus. Int J Audiol. 2025 Oct 4:1-9. doi: 10.1080/14992027.2025.2561889. Online ahead of print. PMID 41046328

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants were assigned to CP1110 Sound Processor System with automated ForwardFocus On (SCAN 2 FF), CP1110 Sound Processor System with ForwardFocus Off (SCAN 2) compared to the previously marketed Nucleus 7 Sound Processor (Model: CP1000).
Period: CP1110 With ForwardFocus On (SCAN 2 FF)
Arm/Group | All Participants
Started | 20
Completed | 20
Not Completed | 0
Period: CP1110 With ForwardFocus Off (SCAN 2)
Arm/Group | All Participants
Started | 20
Completed | 20
Not Completed | 0
Period: CP1000
Arm/Group | All Participants
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants were assigned to CP1110 Sound Processor System with ForwardFocus On (SCAN), CP1110 Sound Processor System with ForwardFocus Off (SCAN) compared to the previously marketed Nucleus 7 Sound Processor (Model: CP1000) in a random order.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 61 [28 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 20
Age of onset of hearing loss [Mean (Standard Deviation); unit: years] | 21.4 (19.84)

OUTCOME MEASURES:

1. Primary Outcome: Speech Reception Thresholds (SRT) Assessed in Spatially Separated Speech and Noise (S0Nrearhalf)
Description: Paired difference in dB SRT (AuSTIN) between the CP1110 Sound Processor with automated ForwardFocus ON (SCAN 2 FF) and ForwardFocus OFF (SCAN 2) in 65 dB SPL S0Nrearhalf 4TB.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: dB SRT
Groups:
- Within-subject Comparison of CP1110 ForwardFocus On Versus ForwardFocus Off in S0Nrearhalf: All participants were assigned to CP1110 Sound Processor System with automated ForwardFocus On (SCAN 2 FF), CP1110 Sound Processor System with ForwardFocus Off (SCAN 2) compared to the previously marketed Nucleus 7 Sound Processor (Model: CP1000). Participants' speech performance (sentences in noise score) in 65 dB SPL S0Nrearhalf 4 Talker Babble was assessed between two programs in CP1110 Sound Processor: automated ForwardFocus On (SCAN 2 FF) versus ForwardFocus Off (SCAN 2).
Arm/Group | Within-subject Comparison of CP1110 ForwardFocus On Versus ForwardFocus Off in S0Nrearhalf
Number analyzed (Participants) | 20
dB SRT
  CP1110 ForwardFocus On | -10.34 [-11.10 to -9.57]
  CP1110 ForwardFocus Off | -6.04 [-7.32 to -4.76]
  Difference between CP1110 ForwardFocus On and ForwardFocus off | -4.30 [-5.19 to -3.41]

2. Secondary Outcome: Speech Reception Thresholds (SRT) Assessed in Spatially Separated Speech and Noise (S0N3)
Description: Paired difference in dB SRT (AuSTIN) between the CP1110 Sound Processor with automated ForwardFocus On (SCAN 2 FF) and ForwardFocus OFF (SCAN 2) in 65 dB SPL S0N3 Babble.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: dB SRT
Groups:
- Within-subject Comparison of CP1110 ForwardFocus On Versus ForwardFocus Off in S0N3: All participants were assigned to CP1110 Sound Processor System with automated ForwardFocus On (SCAN 2 FF), CP1110 Sound Processor System with ForwardFocus Off (SCAN 2) compared to the previously marketed Nucleus 7 Sound Processor (Model: CP1000). Participants' speech performance (sentences in noise score) in 65 dB SPL S0N3 speaker configuration was assessed between two programs in CP1110 Sound Processor: automated ForwardFocus On (SCAN 2 FF) versus ForwardFocus Off (SCAN 2).
Arm/Group | Within-subject Comparison of CP1110 ForwardFocus On Versus ForwardFocus Off in S0N3
Number analyzed (Participants) | 20
dB SRT
  CP1110 ForwardFocus On | -8.35 [-9.68 to -7.01]
  CP1110 ForwardFocus Off | -4.16 [-5.49 to -2.83]
  Difference between CP1110 ForwardFocus On and ForwardFocus Off | -4.18 [-4.90 to -3.47]

3. Secondary Outcome: Adult Cochlear Implant Recipient Speech Perception in Quiet With the CP1110 Sound Processor and the Nucleus 7 Sound Processor
Description: Paired difference in percentage CNC Words correct in quiet (50 dB) with the CP1110 Sound Processor and Nucleus 7 Sound Processor.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: percentage of correct words
Groups:
- Within-subject Comparison of CP1110 Versus Nucleus 7 Sound Processor for Monosyllabic Words in Quiet: All participants underwent a monosyllabic CNC words in quiet test comparing the CP1110 Sound Processor and to the previously marketed Nucleus 7 Sound Processor (Model: CP1000).
Arm/Group | Within-subject Comparison of CP1110 Versus Nucleus 7 Sound Processor for Monosyllabic Words in Quiet
Number analyzed (Participants) | 20
percentage of correct words
  CP1110 Sound Processor | 60.40 [54.81 to 65.99]
  Nucleus 7 Sound Processor | 56.80 [50.37 to 63.23]
  Difference between CP1110 and Nucleus 7 Sound Processor | 3.60 [0.77 to 6.43]

4. Secondary Outcome: Adult Cochlear Implant Subjective Hearing Performance and Sound Quality With the CP1110 Sound Processor and Nucleus 7 Sound Processor
Description: Paired difference in Global Speech, Spatial and Qualities of Hearing Scale (SSQ12) scores after experience with the CP1110 Sound Processor and Nucleus 7 Sound Responses. SSQ12 have a minimum value of 0 and a maximum of 10, wherein a higher score means a better outcome.
Time Frame: Baseline (Nucleus 7) and Visit 2 (6 months, CP1110)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Within-subject Comparison of SSQ12 at Baseline (Nucleus 7) Versus at Visit 2 (CP1110): All 20 participants were assigned to investigate the acceptance and performance of a new behind-the-ear sound processor (Model: CP1110), as compared to the previously marketed Nucleus 7 Sound Processor (Model: CP1000). A key focal point of the investigation was to evaluate the performance of a new implementation of the ForwardFocus noise reduction algorithm in the Automatic Scene Classifier, SCAN 2.
Arm/Group | Within-subject Comparison of SSQ12 at Baseline (Nucleus 7) Versus at Visit 2 (CP1110)
Number analyzed (Participants) | 20
units on a scale
  CP1110 Sound Processor | 5.96 [5.27 to 6.65]
  Nucleus 7 Sound Processor | 5.95 [5.19 to 6.71]
  Difference between CP1100 and Nucleus 7 Sound Processor | 0.01 [-0.58 to 0.61]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- All Participants: All 20 participants were assigned to investigate the acceptance and performance of a new behind-the-ear sound processor (Model: CP1110) with the ForwardFocus feature turned on and off, as compared to the previously marketed Nucleus 7 Sound Processor (Model: CP1000).
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 13/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=20)
Headache (Investigations) | 2 (2) — Headache from CP1110 magnet being too strong.
Bodyache (General disorders) | 1 (1)
Common cold (General disorders) | 1 (1)
Cough (General disorders) | 2 (2)
High fever (General disorders) | 1 (1)
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
One sided headache and neck pain (General disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin lump (Skin and subcutaneous tissue disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Urine retention (Renal and urinary disorders) | 1 (1)
Viral infection (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT05080283/Prot_SAP_000.pdf